CLINICAL TRIAL: NCT01364636
Title: Accuracy of Urinary Neutrophil Gelatinase-Associated Lipocalin (NGAL) in Predicting Cardio-renal Syndrome in Acute Decompensated Heart Failure at Emergency - CYNDERELA-HF Study
Brief Title: Accuracy of Urinary NGAL in Predicting CardioRenal Syndrome in Acute Heart Failure at Emergency - CYNDERELA-HF Study
Acronym: CYNDERELA-HF
Status: Terminated | Type: Observational
Why Stopped: problems with the stability of samples collected
Sponsor: Pro-Cardiaco Hospital (Other)
Collaborators: Universidade Federal Fluminense (Other); Hospital Universitário Antonio Pedro (Other); Diagnósticos da América S.A. (Unknown)
Responsible Party: Evandro Tinoco Mesquita, PhD, Coordinator of Post Graduation Courses of the Department of Cardiovascular Sciences, Fluminense Federal University, Medical Director Hospital PróCardíaco, Department of Cardiovascular Sciences - Fluminense Federal University, Hospital PróCardíaco
Other Study IDs: CYNDERELA-HF
Record Dates: First submitted 2011-05-09; First posted 2011-06-02 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2011-04

CONDITIONS: Cardiorenal Syndrome
Keywords: 1-Heart Failure; 2-Acute Heart Failure; 3-Acute Decompensated Heart Failure; 4-Worsening Renal Function; 5-Acute Kidney Injury; 6-Cardiorenal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine plasma serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Heart Failure: Patients admitted to emergency room in Acute Heart Failure at Hospital PróCardíaco and Hospital Universitario Antonio Pedro

SUMMARY:
Rationale: Heart Failure (HF) elevated prevalence in Brasil and the world; 20-30% AHF patients develop CardioRenal Syndrome (CRS) type 1; Worsening Renal Failure (WRF) is a prognostic marker of mortality in Acute HF;NGAL is a novel biomarker of Acute Kidney Injury released in 2 hours, and addressed in several different clinical scenarios(contrast injury, cardiopulmonary bypass, critical illness.

Hypothesis: Admission NGAL predicts CRS in AHF patients admitted to the Emergency Room (ER).

Primary goal: To evaluate the diagnostic accuracy and the best cutoff value of urinary NGAL to predict the development of CRS type 1 in patients admitted to the Emergency Room.

Secondary goals: 1- To evaluate the prognostic impact of NGAL on in-hospital adverse outcomes (length of hospitalization, death, institution of renal replacement therapy, use of vasoactive drugs, mechanical ventilation).2- Evaluate the prognostic impact of NGAL in adverse outcomes in 30 days, 60 days and 6 months (death, rehospitalization, institution of renal replacement therapy).3- Identify clinical and hemodynamic characteristics of Acute HF that can influence the evolutionary behavior of NGAL levels in 48 hours.4- Identify the association of drugs commonly used for HF management, which might influence the evolutionary behavior of NGAL levels in 48 hours.5-Assess the impact of NGAL results in clinical decision making.

Methods: Observational, prospective, blinded study. Population: Acute HF patients admitted to the ER of Hospital Pró Cardiaco and Hospital Antonio Pedro - Universidade Federal Fluminense.

Statistics: Convenience Sample size (n=180); determination of best cut-off: ROC analysis; Predictive performance of the cut-off: sensibility, specificity, likelihood ratio, predictive value, accuracy; Identification of variables to predict CRS: logistic regression and square-Qui test; Correlations analysis of normally distributed variables: Pearson's linear correlation test; Mean values for normally distributed variables: Mann-Wittney test; Significance on p<0,05; Intra-assay variation analysis.

Study chronogram: Recruitment: 12 months; Results analysis and conclusions: 60 days; Manuscript preparation for paper submission: 30 days.

DETAILED DESCRIPTION:
Rationale: Heart Failure (HF) elevated prevalence in Brasil and the world; 20-30% AHF patients develop CardioRenal Syndrome (CRS) type 1; Worsening Renal Failure (WRF) is a prognostic marker of mortality in Acute HF; available biomarker shows irreversible damage, late in CRS evolution.(creatinine);NGAL is a novel biomarker of Acute Kidney Injury released in 2 hours, and addressed in several different clinical scenarios(contrast injury, cardiopulmonary bypass, critical illness...); Acute HF patient's risk stratification will allow appropriate resource allocation and establishment of criteria for hospital admission and discharge.

Hypothesis: Admission NGAL predicts CRS in AHF patients admitted to the Emergency Room (ER).

Primary goal: To evaluate the diagnostic accuracy and the best cutoff value of urinary NGAL to predict the development of CRS type 1 in patients admitted to the Emergency Room.

Secondary goals: 1- To evaluate the prognostic impact of NGAL on in-hospital adverse outcomes (length of hospitalization, death, institution of renal replacement therapy, use of vasoactive drugs, mechanical ventilation).2- Evaluate the prognostic impact of NGAL in adverse outcomes in 30 days, 60 days and 6 months (death, rehospitalization, institution of renal replacement therapy).3- Identify clinical and hemodynamic characteristics of Acute HF that can influence the evolutionary behavior of NGAL levels in 48 hours.4- Identify the association of drugs commonly used for HF management, which might influence the evolutionary behavior of NGAL levels in 48 hours.5-Assess the impact of NGAL results in clinical decision making.

Methods: Observational, prospective, blinded study. Population: Acute HF patients admitted to the ER of Hospital Pró Cardiaco and Hospital Antonio Pedro - Universidade Federal Fluminense.

Statistics: Convenience Sample size (n=180); determination of best cut-off: ROC analysis; Predictive performance of the cut-off: sensibility, specificity, likelihood ratio, predictive value, accuracy; Identification of variables to predict CRS: logistic regression and square-Qui test; Correlations analysis of normally distributed variables: Pearson's linear correlation test; Mean values for normally distributed variables: Mann-Wittney test; Significance on p<0,05; Intra-assay variation analysis.

Study chronogram: Recruitment: 12 months; Results analysis and conclusions: 60 days; Manuscript preparation for paper submission: 30 days.

ELIGIBILITY:
Inclusion Criteria:

* acute heart failure according to the Framingham's criteria
* informed consent signed

Exclusion Criteria:

* Acute coronary syndrome
* cardiogenic shock
* terminal renal disease
* transplanted patients
* known nephrotoxicity exposure
* urinary tract infection
* sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Emergency rooms of Hospital PróCardíaco and Hospital Universitário Antonio Pedro, presenting with acute heart failure according to the Framingham's criteria. The subjects must sign the informed consent term.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
CardioRenal Syndrome type 1 development | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  CardioRenal Syndrome type 1 development defined by the elevation of serum creatinine of 0,3mg/dL and/or of 50% of baseline values

SECONDARY OUTCOMES:
length of hospitalization | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  number of days of the study entry hospitalization
in-hospital death | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  Death within the study entry hospitalization period
institution of renal replacement therapy | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  need for any kind of dyalisis procedure.
need to use of vasoactive drugs | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  if the patient was submitted to use of vasoactive drugs as dopamine, dobutamine, noradrenaline, milrinone, and other vasoactive drugs
mechanical ventilation | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  if the patient was submitted to mechanical ventilation during the hospitalization period
death | patients will be followed up to 360 days after hospital discharge
  death after study entry hospitalization discharge
rehospitalization | patients will be followed up to 360 days after hospital discharge
  need to be admitted to any hospital after study entry hospitalization discharge
institution of renal replacement therapy | patients will be followed up to 360 days after hospital discharge
  need to be submitted to any dyalisis procedure after study entry hospitalization discharge

CONTACTS AND LOCATIONS:
Overall Officials: Evandro T Mesquita, PhD, Principal Investigator — Fluminense Federal University - Cardiovascular Sciences Department, coordinator of post graduation courses; Hospital PróCardíaco - Medical Director
Locations (1):
- Hospital Universitário Antonio Pedro, Rio de Janeiro, Rio de Janeiro, Brazil